CLINICAL TRIAL: NCT02815501
Title: Thyroid Dysfunction and Obstetric Complications
Acronym: TDOC
Status: Withdrawn | Type: Observational
Why Stopped: Investigator choice
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI11-PR-DESAILLOUD 2
Record Dates: First submitted 2016-06-24; First posted 2016-06-28 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Pregnancy
Keywords: Thyroid dysfunction; obstetric complications
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples for a laboratory work-up and anti-thyroid antibodies.

GROUPS / COHORTS (1):
- women: attending the emergency room and/or hospitalised or followed for: Spontaneous and/or repeated miscarriage Foetal death Pre-eclampsia Retroplacental haematoma Post-partum haemorrhage Premature delivery
  Blood samples
  Interventions: Biological: blood samples

INTERVENTIONS:
Biological: blood samples — for the determination of thyroid hormones (TSH, FT3, FT4 ) and antibodies against the thyroid (anti TPO antibodies and anti thyroglobulin)

SUMMARY:
Obstetric complications are common and can be responsible for maternal and foetal morbidity and mortality. Thyroid dysfunction has been identified as a possible cause of obstetric complications.

Many studies have been conducted to estimate the prevalence and define the nature of obstetric complications observed in patients with thyroid dysfunction. However, women with obstetric complications are not systematically screened for thyroid dysfunction and no published study has evaluated the prevalence of thyroid dysfunction in women with an obstetric complication. As no consensus has been reached concerning systematic screening for thyroid dysfunction in pregnant women, the identification of new high-risk populations could possibly result in a change of clinical practice.

ELIGIBILITY:
Inclusion Criteria:

women attending the emergency room and/or hospitalised or followed for:

* Spontaneous and/or repeated miscarriage
* Foetal death
* Pre-eclampsia
* Retroplacental haematoma
* Post-partum haemorrhage
* Premature delivery
* who consent to participate in the study.
* Assessment of these women will include blood samples for a laboratory work-up and anti-thyroid antibodies.

Exclusion Criteria:

* normal pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women attending the emergency room and/or hospitalised or followed for:
  * Spontaneous and/or repeated miscarriage
  * Foetal death
  * Pre-eclampsia
  * Retroplacental haematoma
  * Post-partum haemorrhage
  * Premature delivery
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2017-10-26 (Actual); Study Completion 2017-10-26 (Actual)

PRIMARY OUTCOMES:
Prevalence of thyroid dysfunction | Day 0
  Estimate the overall and individual prevalence of thyroid dysfunction (hypothyroidism, hyperthyroidism and thyroid autoimmunity) in patients with obstetrical accident

CONTACTS AND LOCATIONS:
Overall Officials: Rachel DESAILLOUD, MD, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France